CLINICAL TRIAL: NCT01691144
Title: Gynecological Cancer Survivors' Views on Follow-up After Cancer Treatment
Brief Title: Follow-up of Gynecological Cancer Patients, Their Needs and Expectations, A Cooperation Project
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Heidi Lidal Fidjeland, MD, University of Oslo
Other Study IDs: 2012/355B
Record Dates: First submitted 2012-08-15; First posted 2012-09-24 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Endometrial Cancer; Ovarian Cancer; Cervical Cancer
Keywords: cancer; gynecological; expectations; satisfaction; cooperation
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Neoplasms; Personal Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- recently treated patients
- 2-3 years after treatment

SUMMARY:
Follow-up of cancer patients accounts for a substantial part of outpatient activity, and alternative models of care are developing. In some countries, low-risk follow-up is already done in primary care, mainly in breast, and colorectal cancer. In this study the investigators will explore gynecological cancer patients about their expectations regarding their future follow-up plan. Further, the investigators will ask about the experience and satisfaction among patients who have already attended a follow-up programme for 2-3 years. In addition, the investigators will especially focus on the cooperation aspect between primary and secondary care. The investigators hypothesize that follow-up of selected gynecological cancer patients can be done by general practitioners.

DETAILED DESCRIPTION:
After gynaecological cancer patients have completed their treatment, they are followed up at a gynaecological outpatient clinic for a number of years. The aim of such follow-up is to detect recurrence, improve survival and reduce adverse effects of the treatment. The national guide for oncological gynaecology recommends follow-up by a specialist for five years at intervals depending on cancer type. Several review studies on follow-up of endometrial, cervical and ovarian cancer patients show large international variations in follow-up routines. There are only retrospective studies available, and they indicate that most recurrences are discovered within the first three years after completed treatment, and, in most cases, by the women themselves. More intensive surveillance does not appear to affect the time for discovery of recurrence.

A few randomised controlled studies and retrospective cohort studies have been published that focus on follow-up of colon cancer and breast cancer patients by general practitioners versus by hospital specialists. These studies have not shown any significant differences between the groups in terms of detection of recurrence, incidence of serious clinical events connected with recurrence or health-related quality of life.

The investigators therefore plan to perform a study in which both gynaecological cancer patients and their regular general practitioners are asked about their views on patient follow-up after completed treatment. The investigators especially wish to focus on the collaboration aspect.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* histologically or cytologically proven cancer

Exclusion Criteria:

* Unability to fill out questionnaires (due to language or cognitive barriers)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly treated gynecological cancer patients and patients treated 2-3 years ago
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Patient expectation questionnaire | within the first 30 days after primary treatment
  The patients will be asked to fill in a quesionnaire regarding their expectations on follow-up care

SECONDARY OUTCOMES:
Patient satisfaction questionnaire | 3 years after treatment
  The patients will be asked to fill in a quesionnaire regarding their satisfaction on follow-up care after three years

CONTACTS AND LOCATIONS:
Overall Officials: Mette Brekke, PhD, Study Chair — University of Oslo
Locations (2):
- Norway (2):
  - Sorlandet Hospital Kristiansand, Kristiansand
  - St. Olavs Hospital, Trondheim

REFERENCES:
- [Background] Vistad I, Moy BW, Salvesen HB, Liavaag AH. Follow-up routines in gynecological cancer - time for a change? Acta Obstet Gynecol Scand. 2011 Jul;90(7):707-18. doi: 10.1111/j.1600-0412.2011.01123.x. Epub 2011 Apr 15. PMID 21382018
- [Background] Vistad I, Cvancarova M, Salvesen HB. Follow-up of gynecological cancer patients after treatment - the views of European experts in gynecologic oncology. Acta Obstet Gynecol Scand. 2012 Nov;91(11):1286-92. doi: 10.1111/j.1600-0412.2012.01523.x. Epub 2012 Sep 18. PMID 22880840